CLINICAL TRIAL: NCT03602794
Title: A Comparison of Local Infiltration Analgesia and Pecs Block for Analgesia in Mastectomy With Axillary Dissection - an Equivalence Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Louis Ng Xiang Long (Other)
Responsible Party: Sponsor-Investigator, Louis Ng Xiang Long, Co- Investigator, Changi General Hospital
Organization: Changi General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2017/2894
Record Dates: First submitted 2018-07-18; First posted 2018-07-27 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Mastectomy; Lymphedema; Local Infiltration; Anesthesia, Local; Block
MeSH Terms: conditions — Lymphedema; Bites and Stings | interventions — Anesthesia, Local

STUDY DESIGN:
Intervention Model Description: Randomised Controlled
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PECs Block (Active Comparator): Total local anaesthetic dose: 30ml ropivacaine 0.5%
  •Pecs block will be performed by anaesthetist using ultrasound guidance in plane approach: 10ml ropivacaine 0.5% will be delivered at the plane between pectoralis major and pectoralis minor, another 20ml ropivacaine 0.5% will be delivered in the plane between the pectoralis minor and serratus anterior muscles at the level of the third and fourth ribs
  Interventions: Procedure: PECs Block
- Local Infiltration (Placebo Comparator): LIA will be performed by surgeon during the operation. The upper skin flap will be raised in the standard manner for mastectomy. The lateral border of the major pectoralis muscle will then be visualised. A volume of 10 ml ropivacaine 0.5% will be delivered between the inter-fascial planes of the pectoral muscles. The lower skin flap will then be raised in the standard manner for mastectomy and the breast is raised off the pectoralis muscle exposing the serratus anterior muscle. A volume of 20 ml ropivacaine 0.5% will be delivered between the muscle planes of the serratus anterior and pectoralis minor muscles.
  Interventions: Procedure: Local infiltration

INTERVENTIONS:
Procedure: PECs Block — Regional Anaesthesia Technique ie Pectoralis Nerve Block under ultrasound guidance
  Arms: PECs Block
Procedure: Local infiltration — LIA will be performed by surgeon during the operation. The upper skin flap will be raised in the standard manner for mastectomy. The lateral border of the major pectoralis muscle will then be visualised. A volume of 10 ml ropivacaine 0.5% will be delivered between the inter-fascial planes of the pectoral muscles. The lower skin flap will then be raised in the standard manner for mastectomy and the breast is raised off the pectoralis muscle exposing the serratus anterior muscle. A volume of 20 ml ropivacaine 0.5% will be delivered between the muscle planes of the serratus anterior and pectoralis minor muscles.
  Arms: Local Infiltration

SUMMARY:
The investigators aim to compare the quality of pain relief provided by local infiltration analgesia delivered by surgeon and Pecs block delivered by anaesthetist under ultrasound guidance for patients undergoing mastectomy with axillary dissection.

DETAILED DESCRIPTION:
Total breast removal with armpit dissection may be a painful surgery. Pectoral nerve block (Pecs block) is common pain relief method used to reduce pain after breast surgery.

The Pecs block is a pain relief method technique at targeted body part. The Pecs block numbs nerves which supply sensation to the upper chest wall, armpit and upper arm. This procedure is only possible under ultrasound guidance and is carried out by the anaesthetist (medical specialist who administers anaesthetics) after patients are put under general anaesthesia.

Despite the advantages of Pecs block in pain management, this method is not always available to all patients due to various reasons. These reasons include the availability of ultrasound machine to facilitate the method, presence of anaesthetist to carry out the procedure and additional time required to perform this method in the operating theatre.

Another method has been modified by our surgeons (medical specialist who performs surgery, a different specialty from anaesthetist) to achieve pain relief among patients undergoing breast removal surgery. This method is called local infiltration analgesia (LIA). The pain control is achieved by having the surgeons to deliver a pain control drug surgically during the breast removal operation. LIA could be a good pain control alternative when a Pecs block could not be performed.

The investigators hope to compare the quality of pain relief provided by local infiltration analgesia delivered by surgeon and Pecs block delivered by anaesthetist under ultrasound guidance. The investigators hope to show that LIA delivered by surgeon is as effective as Pecs block in patients undergoing mastectomy with axillary dissection.

ELIGIBILITY:
Inclusion Criteria:

* Age above 21 years old
* Able to give consent
* Body weight > 50kg

Exclusion Criteria:

* Patient's refusal and inability to give consent
* Allergy or contraindicated to local anaesthetics, paracetamol, NSAIDS or opioids
* Background history of chronic pain
* Bilateral procedures

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 40 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-07-16 (Estimated); Study Completion 2019-07-16 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption in 24 hour after surgery | 24 hour
  Total morphine consumption in 24 hour after surgery

SECONDARY OUTCOMES:
Duration of analgesia | 24 hours
  time to first rescue analgesia after administration of block
Postoperative pain score. | 24 hours
  Post op pain score will be assessed using a visual analogue scale (VAS, 0-10; 0 = no pain and 10 = worst imaginable pain). The vital signs and pain score will be recorded at 0, 0.5, 1, 2, 4, 6, 8, 12, and 24 h after surgery by the attending staff nurses blinded to the group allocation
Adverse Effects | 24 hours
  Any adverse effects will be recorded (such as hypotension, respiratory depression, pruritus, shivering and urinary retention)
Postoperative nausea vomiting (PONV) | 24 hours
  Postoperative nausea vomiting (PONV)
Intraoperative analgesia | 24 hours
  total usage of IV Fentanyl intraoperatively
Operative time | 24 hrs
  duration of surgery
Block performance time | 24 hours
  time from needle insertion until needle exit from the skin
Block related complications | 24 hours
  pneumothorax
Block related complications | 24 hours
  vascular puncture
Block related complications | 24 hours
  local anaesthetic toxicity
Post-operative complications | 24 hours
  Bleeding
Post-operative complications | 24 hours
  Wound infection

CONTACTS AND LOCATIONS:
Overall Officials: Kwee Lian Woon, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blanco R, Fajardo M, Parras Maldonado T. Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):470-5. doi: 10.1016/j.redar.2012.07.003. Epub 2012 Aug 29. PMID 22939099
- See also: Ultrasound description of Pecs II (modified Pecs I): A novel approacj to breast surgery — http://dx.doi.org/10.1016/j.redar.2012.07.003